CLINICAL TRIAL: NCT04308811
Title: Platelet-Rich Plasma in the Management of Asherman Syndrome
Brief Title: Autologous Platelet-Rich Plasma in the Management of Asherman Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed I Amer, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASU456
Record Dates: First submitted 2018-12-14; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Intervention Model Description: The patients who are diagnosed previously with severe AS will choose an envelope which determines the treatment method. There will be 60 envelops assigning for the groups mixed together in one box. This will ensure a randomized allocation of patients to either group of this study. Hysteroscopy adhesiolysis will be done to all participants in the study. in the first group, Adhesiolysis will be followed by intrauterine use of PRP then insertion of Foley balloon catheter. in the second group, adhesiolysis will be followed by insertion of Foley balloon catheter covered by freeze-dried amniotic graft. In the third group, Adhesiolysis will be followed by insertion of Foley balloon catheter. All foley ballon removed 2 weeks postoperative. All patients will be given antibiotics and hormonal treatment. Also, they will be given low dose aspirin and sildenafil 50mg daily.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- platelet rich plasma group (Other): intrauterine platelet rich plasma injection and intrauterine balloon insertion after hysteroscopic lysis of intrauterine adhesions
  Interventions: Biological: platelet rich plasma
- amniotic membrane graft group (Other): the clinician will perform hysteroscopic lysis of intrauterine adhesions followed by application of intrauterine balloon covered by freeze-dried amniotic membranes.
  Interventions: Combination Product: amniotic membrane graft group
- intrauterine balloon group (Other): the clinician will perform hysteroscopic lysis of intrauterine adhesions followed by application of intrauterine balloon
  Interventions: Device: Intrauterine balloon

INTERVENTIONS:
Biological: platelet rich plasma — Platelet rich plasma and intrauterine balloon applied intrauterine after hysteroscopic adhesiolysis of intrauterine adhesions
  Arms: platelet rich plasma group
Combination Product: amniotic membrane graft group — amniotic membrane applied on the intrauterine balloon after hysteroscopic lysis of intrauterine adhesions
  Arms: amniotic membrane graft group
Device: Intrauterine balloon — intrauterine balloon applied intrauterine after hysteroscopic lysis of intrauterine adhesions
  Arms: intrauterine balloon group

SUMMARY:
The aim of the study is to find out the benefit of the platelet-rich plasma in preventing reformation of intrauterine adhesions after adhesiolysis in cases of Asherman syndrome

DETAILED DESCRIPTION:
Patients fulfilling criteria will be randomized into three equal groups. The patients who are diagnosed previously with severe AS will choose an envelope which determines the treatment method. There will be 60 envelops assigning for the groups mixed together in one box. This will ensure a randomized allocation of patients to either group of this study.

Hysteroscopy adhesiolysis will be done to all participants in the study. in the first group, Adhesiolysis will be followed by intrauterine use of PRP then insertion of intrauterine Foley balloon catheter that will be inflated and left for 2 weeks. in the second group, adhesiolysis will be followed by insertion of intrauterine Foley balloon catheter covered by freeze-dried amniotic graft and will be inflated and left for 2 weeks. In the third group, Adhesiolysis will be followed by insertion of intrauterine Foley balloon catheter that will be inflated and left for 2 weeks. All patients will be given antibiotics and hormonal treatment. Also, they will be given low dose aspirin and sildenafil 50mg daily.

ELIGIBILITY:
Inclusion Criteria: Severe intrauterine synechia confirmed by hysteroscopy

* age group from 20 to 40 years

Exclusion Criteria:

* Hemoglobin less than 11 g/dl
* Platelet less than 150000/mm3
* Patients taking anticoagulants
* Patients taking NSAID in the 15 days prior to the procedure
* Active cervical or uterine infection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Grade of intrauterine adhesions | after one month
  Grade of intrauterine adhesions

SECONDARY OUTCOMES:
menstruation | within three months postoperative
  amount of menstrual blood change

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy unit, Ain shams university Maternity hospital, Cairo, Egypt